CLINICAL TRIAL: NCT00229424
Title: Verification Study on Lafutidine in Mild Reflux Oesophagitis - Double Blind Controlled Study With Famotidine -
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Taiho Pharmaceutical Co., Ltd., Taiho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10019350; LAF/GER/3D1/FN/01
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Gastroesophageal Reflux
Keywords: lafutidine; reflux oesophagitis; Gastroesophageal Reflux; famotidine; Double Blind; Controlled Study; H2 receptor antagonist; H2-blocker
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis, Peptic | interventions — lafutidine; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Lafutidine group
  Interventions: Drug: Lafutidine
- 2 (Active Comparator): Famotidine group
  Interventions: Drug: Famotidine
- 3 (Placebo Comparator): Placebo group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lafutidine — Oral administration of lafutidine by 20mg/day along with famotidine placebo
  Arms: 1
Drug: Famotidine — Oral administration of famotidine by 40mg/day along with lafutidine placebo
  Arms: 2
Other: Placebo — Oral administration of lafutidine placebo along with famotidine placebo
  Arms: 3

SUMMARY:
The purpose of the study is to verify superiority of the lafutidine group over the placebo group and non-inferiority to the famotidine group in terms of endoscopic healing rate of the patients with mild reflux oesophagitis.

Furthermore, the followings are compared:

The improvement effect in heartburn and other subjective symptoms, and dosing frequency of MALFA ® suspension (neutralizer) as well as incidence of adverse events among the lafutidine 20 mg/day treatment group, the famotidine 40 mg/day treatment group and the placebo treatment group in patients with mild reflux oesophagitis.

DETAILED DESCRIPTION:
In Japan it is reported that many patients with reflux oesophagitis are relatively mild and do not usually require strong treatment, and even H2 receptor antagonists are considered to demonstrate sufficient healing effects. Haruma thinks that the first choice should be PPI in principle which has the best therapeutic effect as the medical guideline if a patient has a strong reflux symptom such as heartburn or is diagnosed with severe reflux oesophagitis (Grade C or D according to the Los Angels Classification) as a result of the upper gastrointestinal endoscopic test. Later, after healing is confirmed at 8 weeks of treatment or after the subjective symptoms have been improved, the dose of PPI should be reduced to half to transfer to maintenance therapy. On the other hand, if a patient has mild subjective symptoms or develops mild reflux oesophagitis (Grade A or B according to the Los Angels Classification) as a result of the upper gastrointestinal endoscopic test, only about 10% of such patients aggravate in the long-run and some patients heal in the natural course. Therefore, considering that Japanese gastric-acid secretion is lower than Westerners, they recommend that antacids such as H2 receptor antagonists or sodium alginates is used to treat symptoms as they appear along with the improvement in the lifestyle. As mentioned above, lafutidine that strongly suppresses acid secretion during the daytime from the initial phase of treatment is expected to demonstrate sufficient effect in treatment of mild reflux oesophagitis similar to the conventional H2 receptor antagonists.

Based on above, the clinical trial is planned with the objective to confirmedly demonstrate the efficacy of lafutidine in mild reflux oesophagitis.

Comparisons: The endoscopic healing rate of lafutidine in the patients with mild reflux oesophagitis is compared to the rate of placebo and it is also compared to the rate of famotidine.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 and over (at the time of consent given)
* Gender and inpatient or outpatient: Irrelevant
* Patients diagnosed with Grade A or Grade B mild reflux oesophagitis (according to the Los Angels classification) through endoscopic test
* Patients who complained about "heartburn symptom" within one week prior to the enrollment

Exclusion Criteria:

* Patients whose "heartburn symptom" has been disappeared (not been observed at all) during the observation period (Check before official enrollment)
* Patients in ill compliance with dosing the investigational product for the observation period (Not more than 75%, check from the patient dairy before official enrollment)
* Patients the investigator/sub-investigator assessed difficult to complete the patient diary during the treatment period because the patient diary for the observation period has too many deficiencies. (Check before official enrollment)
* Patients with complication of gastric/duodenal ulcer (scarring acceptable)
* Patients with complication of Barrett lining over the site exceeding 3 cm of esophageal distal portion
* Patients who have received the normal dose of H2 receptor antagonist or proton pump inhibitor (PPI) for 8 weeks in vain
* Patients whose Helicobacter pylori was successfully eradicated within 24 weeks
* Patients with medical history of upper gastrointestinal tract excision
* Patients with complication of angina pectoris
* Patients who have received treatment of any other investigational product within 12 weeks
* Patients who showed any of the following values at the laboratory tests before official enrollment: Hemoglobin: < 9.5 g/dL, WBC: < 3,000/mm^3, Thrombocytes: < 75,000/mm^3, AST and ALT : ≥ 100 IU/L, Creatinine: ≥ 1.5 mg/dL These should be assessed using the current test values from the blood drawn within 4 weeks prior to official enrollment.
* Patients with complication of serious cardiac disorder (Grade 3 or above under PAB/SD Notification No. 80) For example, patients with triplet or more ventricular premature contractions (multi-sources) or using a pacemaker
* Patients with medical history of serious hypersensitivity to drugs (Grade 3 or above under PAB/SD Notification No. 80)
* Patients who receive treatment of cancer
* Women of confirmed or potential pregnancy, those who wish to become pregnant, and breast feeding women
* Patients having any other condition that, in the opinion of the investigator/sub-investigator disqualifies them for the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325
Dates: Start 2005-04; Primary Completion 2006-10 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Endoscopic healing rate | At the eighth week after treatment

SECONDARY OUTCOMES:
Frequency of heartburn symptom, intensity and improvement effect in other subjective symptoms and dosing frequency of MALFA ® suspension (neutralizer) | Everyday

CONTACTS AND LOCATIONS:
Overall Officials: Tomoyuki Koike, MD, Principal Investigator — Tohoku University Hospital
Locations (1):
- Tohoku University Hospital, 1-1, Seiryo-cho, Aoba-ku, Sendai, Miyagi, Japan

REFERENCES:
- [Result] Ohara S, Haruma K, Kinoshita Y, Kusano M. [Efficacy evaluation of lafutidine for mild reflux esophagitis in Japanese patients]. Nihon Shokakibyo Gakkai Zasshi. 2010 Apr;107(4):588-97. Japanese. PMID 20379093